CLINICAL TRIAL: NCT01515423
Title: A Randomized, Multicenter, Double-Blind, Non-inferiority Study of Paliperidone Palmitate 3 Month and 1 Month Formulations for the Treatment of Subjects With Schizophrenia
Brief Title: Study of Paliperidone Palmitate 3 Month and 1 Month Formulations for the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100662; R092670PSY3011 (Other: Janssen Research & Development, LLC); 2011-004889-15 (EudraCT Number); U1111-1135-7054 (Other: Universal Trial Number)
Record Dates: First submitted 2012-01-17; First posted 2012-01-24 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; R092670; Paliperidone Palmitate; Paliperidone palmitate 1 month formulation (PP1M); Paliperidone palmitate 3 month formulation (PP3M)
MeSH Terms: conditions — Schizophrenia | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone palmitate 3-month (PP3M) (Experimental): A formulation of paliperidone palmitate with a 3-month injection interval
  Interventions: Drug: PP3M 175 mg eq.; Drug: PP3M 263 mg eq.; Drug: PP3M 350 mg eq.; Drug: PP3M 525 mg eq.; Drug: Placebo (20% Intralipid)
- Paliperidone palmitate 1-month (PP1M) (Active Comparator): A formulation of paliperidone palmitate with a 1-month injection interval
  Interventions: Drug: PP1M 50 mg eq.; Drug: PP1M 75 mg eq.; Drug: PP1M 100 mg eq.; Drug: PP1M 150 mg eq.

INTERVENTIONS:
Drug: PP3M 175 mg eq. — Type= exact number, unit= mg eq., number= 175, form= injection, route= intramuscular use. One injection every third month for 48 weeks.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: PP3M 263 mg eq. — Type= exact number, unit= mg eq., number= 263, form= injection, route= intramuscular use. One injection every third month for 48 weeks.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: PP3M 350 mg eq. — Type= exact number, unit= mg eq., number= 350, form= injection, route= intramuscular use. One injection every third month for 48 weeks.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: PP3M 525 mg eq. — Type= exact number, unit= mg eq., number= 525, form= injection, route= intramuscular use. One injection every third month for 48 weeks.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: Placebo (20% Intralipid) — Form= injection, route= intramuscular use. One injection monthly when not receiving active medication for 48 weeks.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: PP1M 50 mg eq. — Type= exact number, unit= mg eq., number= 50, form= injection, route= intramuscular use. One injection every month for 48 weeks.
  Arms: Paliperidone palmitate 1-month (PP1M)
Drug: PP1M 75 mg eq. — Type= exact number, unit= mg eq., number= 75, form= injection, route= intramuscular use. One injection every month for 48 weeks.
  Arms: Paliperidone palmitate 1-month (PP1M)
Drug: PP1M 100 mg eq. — Type= exact number, unit= mg eq., number= 100, form= injection, route= intramuscular use. One injection every month for 48 weeks.
  Arms: Paliperidone palmitate 1-month (PP1M)
Drug: PP1M 150 mg eq. — Type= exact number, unit= mg eq., number= 150, form= injection, route= intramuscular use. One injection every month for 48 weeks.
  Arms: Paliperidone palmitate 1-month (PP1M)

SUMMARY:
The purpose of this study is to demonstrate that a paliperidone palmitate 3 month formulation (PP3M) is as effective as the paliperidone palmitate 1 month formulation (PP1M) in the treatment of patients with schizophrenia who have been stabilized on PP1M.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), double blind (neither physician nor patient knows the treatment that the patient receives), parallel group (each group of patients will be treated at the same time), multicenter non-inferiority (the effect of the new treatment is not worse than that of the comparison treatment) study. A new formulation of paliperidone palmitate with a 3-month injection interval (PP3M) is being tested for use as maintenance treatment for subjects with schizophrenia who have been first stabilized on paliperidone palmitate with a 1-month injection interval (PP1M). The study consists of 3 phases: a screening/washout/tolerability phase (up to 21 days); a 17-week open-label (all people know the identity of the intervention) stabilization phase (referred to as the Open-label Phase) and a 48-week fixed dose, randomized, double-blind controlled phase (referred to as the Double-blind Phase). After completion of the Screening Phase, all patients will receive PP1M in the Open-label Phase. During this time, flexible dosing will occur at Weeks 5 and 9. At Week 13 patients are to receive the dose of PP1M that was administered at Week 9. Patients who are clinically stable at the end of the Open-label Phase will enter the Double-blind Phase and will be randomly assigned in a 1:1 ratio to receive fixed doses of PP3M or PP1M.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia for more than 1 year and whose symptoms are worsening in the opinion of the investigator
* A total score in the Positive and Negative Syndrome Scale (PANSS) between 70 and 120
* Signed informed consent
* Women must not be pregnant, breastfeeding, and if capable of pregnancy must practice an effective method of birth control
* Men must agree to use a double-barrier method of birth control
* Be medically stable on the basis of clinical laboratory tests, physical examination, medical history, vital signs, and electrocardiogram (ECG)

Exclusion Criteria:

* A diagnosis other than schizophrenia, e.g., dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, schizophreniform disorder, autistic disorder, primary substance-induced psychotic disorder, dementia-related psychosis
* Relevant history or current presence of any significant or unstable medical condition(s) determined to be clinically significant by the Investigator (ie, obesity, diabetes, heart disease etc)
* A diagnosis of substance dependence within 6 months before screening
* History of neuroleptic malignant syndrome (NMS) or tardive dyskinesia
* Clozapine use in the last 2 months when used for treatment-resistant or treatment-refractory illness
* Clinically significant findings in biochemistry, hematology, ECG or urinalysis results
* Any other disease or condition that, in the opinion of the investigator, would make participation not in the best interest of the patient or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1429 (Actual)
Dates: Start 2012-05; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (174):
- United States (24):
  - Little Rock, Arkansas
  - Glendale, California
  - Long Beach, California
  - Oakland, California
  - Oceanside, California
  - Orange, California
  - San Diego, California
  - New Britain, Connecticut
  - Bradenton, Florida
  - Kissimmee, Florida
  - Tampa, Florida
  - Wichita, Kansas
  - East Lansing, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Jamaica, New York
  - Durham, North Carolina
  - Canton, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Bothell, Washington
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Rosario
- Australia (2):
  - Elizabeth Vale
  - Frankston
- Innsbruck, Austria
- Belgium (7):
  - Assebroek
  - Bertrix
  - Dave
  - Heusden
  - Jette
  - Marchienne-au-Pont
  - Sint-Denijs-Westrem
- Rio de Janeiro, Brazil
- Bulgaria (4):
  - Burgas
  - Kazanlak
  - Radnevo
  - Sofia
- Canada (4):
  - Calgary, Alberta
  - Halifax, Ontario
  - Montreal, Quebec
  - Burlington
- China (11):
  - Baoding
  - Beijing
  - Changsha
  - Guangdong
  - Guangzhou
  - Hangzhou
  - Kunming
  - Shanghai
  - Tianjin
  - Wuhan
  - Xi'an
- Czechia (5):
  - Brno
  - Hořovice
  - Liberec
  - Prague
  - Přerov
- France (4):
  - Clermont-Ferrand
  - Dole
  - Montpellier
  - Toulon
- Germany (5):
  - Bochum
  - Gelsenkirchen
  - Hamburg
  - Heidelberg
  - München
- Greece (3):
  - Arta
  - Athens
  - Katerini
- Hungary (5):
  - Balassagyarmat
  - Budapest
  - Gyõr
  - Kalocsa
  - Sopron
- Japan (39):
  - Aizu-Wakamatsu
  - Fujioka
  - Fujisawa
  - Hadano
  - Himeji
  - Hitachi
  - Ichikawa
  - Kanuma
  - Kanzaki
  - Kashihara
  - Kashiwara
  - Kasuya
  - Kawasaki
  - Kitagunma
  - Kochi
  - Kodaira
  - Kumagaya
  - Kumamoto
  - Kure
  - Matsusaka
  - Mitaka
  - Moriguchi
  - Nagasaki
  - Naha
  - Nirasaki
  - Ohta
  - Okayama
  - Okinawa
  - Sakai
  - Shibukawa
  - Takatsuki
  - Toki
  - Tokushima
  - Tokyo
  - Toyoake
  - Ueda
  - Yatsushiro
  - Yokkaichi
  - Yokohama
- Mexico (3):
  - Guadalajara
  - Monterrey
  - Tlalnepantla
- Poland (9):
  - Bełchatów
  - Bydgoszcz
  - Chełmno
  - Gdynia Na
  - Lubin
  - Lubliniec
  - Piekary Śląskie
  - Torun
  - Ząbki
- Portugal (5):
  - Almada
  - Angra do Heroísmo
  - Coimbra
  - Lisbon
  - Porto
- Romania (2):
  - Brasov
  - Cluj-Napoca
- Russia (13):
  - Arkhangelsk
  - Gatchina
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Smolensk Region N/A
  - St-Peterburg
  - Tomsk Na
  - Yaroslavl
  - Yekaterinburg
- Slovakia (4):
  - Bratislava
  - Michalovce
  - Rimavská Sobota
  - Trenčín
- South Korea (4):
  - Busan
  - Gwangju
  - Gyeonggi-do
  - Seoul
- Spain (7):
  - Alicante
  - Barakaldo
  - Barcelona
  - Coslada
  - Elche
  - Madrid
  - Zamora
- Uppsala, Sweden
- Taiwan (3):
  - Bali Township, Taipei County
  - Kaohsiung City
  - Taoyuan District
- Ukraine (5):
  - Hlevakha
  - Kharkiv
  - Kiev
  - Odesa
  - Poltava

REFERENCES:
- [Derived] Li X, Ye C, Zhang W, Jia M, Wang G. Factors Associated with Symptom Stabilization that Allow for Successful Transition from Once-Monthly Paliperidone Palmitate to Three-Monthly Paliperidone Palmitate: A Post Hoc Analysis Examined Clinical Characteristics in Chinese Patients with Schizophrenia. CNS Drugs. 2024 Jan;38(1):55-65. doi: 10.1007/s40263-023-01056-x. Epub 2024 Jan 8. PMID 38190077
- [Derived] Gopal S, Gogate J, Pungor K, Kim E, Singh A, Mathews M. Improvement of Negative Symptoms in Schizophrenia with Paliperidone Palmitate 1-Month and 3-Month Long-Acting Injectables: Results from a Phase 3 Non-Inferiority Study. Neuropsychiatr Dis Treat. 2020 Mar 6;16:681-690. doi: 10.2147/NDT.S226296. eCollection 2020. PMID 32184607
- [Derived] Savitz AJ, Xu H, Gopal S, Nuamah I, Mathews M, Soares B. Efficacy and safety of paliperidone palmitate 3-month formulation in Latin American patients with schizophrenia: A subgroup analysis of data from two large phase 3 randomized, double-blind studies. Braz J Psychiatry. 2019 Nov-Dec;41(6):499-510. doi: 10.1590/1516-4446-2018-0153. PMID 30994855
- [Derived] Nash AI, Turkoz I, Savitz AJ, Mathews M, Kim E. Predictors of achieving remission in schizophrenia patients treated with paliperidone palmitate 3-month formulation. Neuropsychiatr Dis Treat. 2019 Mar 22;15:731-737. doi: 10.2147/NDT.S194264. eCollection 2019. PMID 30962688
- [Derived] Mathews M, Pei H, Savitz A, Nuamah I, Hough D, Alphs L, Gopal S. Paliperidone Palmitate 3-Monthly Versus 1-Monthly Injectable in Patients With Schizophrenia With or Without Prior Exposure to Oral Risperidone or Paliperidone: A Post Hoc, Subgroup Analysis. Clin Drug Investig. 2018 Aug;38(8):695-702. doi: 10.1007/s40261-018-0647-z. PMID 29882073
- [Derived] Magnusson MO, Samtani MN, Plan EL, Jonsson EN, Rossenu S, Vermeulen A, Russu A. Population Pharmacokinetics of a Novel Once-Every 3 Months Intramuscular Formulation of Paliperidone Palmitate in Patients with Schizophrenia. Clin Pharmacokinet. 2017 Apr;56(4):421-433. doi: 10.1007/s40262-016-0459-3. PMID 27743205
- [Derived] Samtani MN, Nandy P, Ravenstijn P, Remmerie B, Vermeulen A, Russu A, D'hoore P, Baum EZ, Savitz A, Gopal S, Hough D. Prospective dose selection and acceleration of paliperidone palmitate 3-month formulation development using a pharmacometric bridging strategy. Br J Clin Pharmacol. 2016 Nov;82(5):1364-1370. doi: 10.1111/bcp.13050. Epub 2016 Jul 24. PMID 27333588

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1429 participants received at least 1 dose of the study agent in the Open-label Phase, out of which 1016 participants were randomized into the Double blind Phase (Safety population).
Groups:
- Open-Label: Paliperidone Palmitate (PP1M) 1-month Formulation: Participants received Paliperidone Palmitate 1-month formulation (PP1M) in a dose of 150 milligram equivalent (mg eq.) on Day 1 and 100 mg eq. on Day 8, both as an injection in the deltoid muscle. The injections at Week 5 (Day 36) and Week 9 (Day 64) given in either the deltoid or gluteal muscle and were flexibly dosed (50, 75, 100, or 150 mg eq.). At Week 13 (Day 92) participants received the same dose of PP1M that was administered at Week 9.
- Double-Blind: Paliperidone Palmitate(PP3M) 3-month Formulation: Participants received Paliperidone Palmitate 3-month formulation (PP3M) in a fixed dose of 3.5 fold multiple of the PP1M dose administered at Week 13, that is participants received fixed dose injections of PP3M (175, 263, 350, or 525 mg eq.) on Week 17, 29, 41, and 53 as injection in deltoid muscle or gluteal muscle.
- Double-Blind: Paliperidone Palmitate(PP1M) 1-month Formulation: Participants received Paliperidone Palmitate 1-month formulation (PP1M) in a fixed dose that was administered at Week 9 at every month for 48 weeks, that is, participants received fixed dose injections of PP1M (50, 75, 100, or 150 mg eq.) as injection on deltoid muscle or gluteal muscle.
Period: Open Label Phase
Arm/Group | Open-Label: Paliperidone Palmitate (PP1M) 1-month Formulation | Double-Blind: Paliperidone Palmitate(PP3M) 3-month Formulation | Double-Blind: Paliperidone Palmitate(PP1M) 1-month Formulation
Started | 1429 | 0 | 0
Completed | 1016 | 0 | 0
Not Completed | 413 | 0 | 0
Not completed — Adverse Event | 57 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Lack of Efficacy | 117 | 0 | 0
Not completed — Lost to Follow-up | 21 | 0 | 0
Not completed — Withdrawal by Subject | 118 | 0 | 0
Not completed — excluded from DB Phase | 70 | 0 | 0
Not completed — Other | 28 | 0 | 0
Period: DOUBLE BLIND
Arm/Group | Open-Label: Paliperidone Palmitate (PP1M) 1-month Formulation | Double-Blind: Paliperidone Palmitate(PP3M) 3-month Formulation | Double-Blind: Paliperidone Palmitate(PP1M) 1-month Formulation
Started | 0 | 504 | 512
Completed | 0 | 422 | 420
Not Completed | 0 | 82 | 92
Not completed — Adverse Event | 0 | 15 | 13
Not completed — Death | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 7 | 12
Not completed — Pregnancy | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 50 | 53
Not completed — Other | 0 | 6 | 12
Not completed — Blind broken by investigator | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomly assigned to treatment during the Double-blind Phase and received at least 1 dose study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind: Paliperidone Palmitate(PP3M) 3-month Formulation | Double-Blind: Paliperidone Palmitate(PP1M) 1-month Formulation | Total
Number analyzed (Participants) | 504 | 512 | 1016
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11.89) | 38.3 (12.24) | 38.6 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 231 | 477
  Male | 258 | 281 | 539
Region of Enrollment [Number; unit: participants]
  China | 104 | 106 | 210
  Russian Federation | 75 | 75 | 150
  Japan | 52 | 56 | 108
  United States | 41 | 48 | 89
  Ukraine | 35 | 29 | 64
  Czech Republic | 31 | 29 | 60
  Hungary | 21 | 19 | 40
  Poland | 17 | 20 | 37
  Argentina | 14 | 16 | 30
  Bulgaria | 12 | 16 | 28
  Brazil | 13 | 12 | 25
  Spain | 11 | 14 | 25
  Slovakia | 12 | 10 | 22
  Portugal | 11 | 10 | 21
  Mexico | 7 | 9 | 16
  Taiwan | 7 | 7 | 14
  Romania | 7 | 6 | 13
  Germany | 8 | 4 | 12
  South Korea | 7 | 5 | 12
  Belgium | 7 | 4 | 11
  Greece | 5 | 6 | 11
  Canada | 3 | 6 | 9
  Australia | 3 | 2 | 5
  France | 1 | 2 | 3
  Austria | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Relapse at Week 48 During the Double-Blind Phase
Description: Relapse defined as: Psychiatric hospitalization;participant had an increase of 25 percent in total PANSS score from randomization for 2 consecutive assessments separated by 3-7 days if score at randomization was greater than (>) 40; had a 10 point increase in total PANSS score from randomization for 2 consecutive assessments separated by 3-7 days if score at randomization was less than or equal to (<=) 40; deliberate self-injury or exhibited violent behavior resulting in suicide, clinically significant injury;suicidal or homicidal ideation and aggressive behavior;For PANSS items-had a score of greater than or equal to (>=) 5 after randomization for 2 consecutive assessments separated by 3-7 days on any of above items if maximum score for these above PANSS items was <=3 at randomization; had a score of >=6 after randomization for 2 consecutive assessments separated by 3-7 days on any of above items if maximum score for these above PANSS items was 4 at randomization.
Time Frame: Up to 48 weeks
Population: Modified intent-to-treat (mITT) analysis set included all participants who were randomly assigned to treatment during Double-blind Phase, received at least 1 dose of study drug and did not have any errors in delivery of active treatment. Here,N=number of participants analysed is the total participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Groups:
- Double Blind: Paliperidone Palmitate 3 Month Formulation: Participants received Paliperidone Palmitate 3-month formulation (PP3M) in a fixed dose of 3.5 fold multiple of the PP1M dose administered at Week 13, that is participants received fixed dose injections of PP3M (175, 263, 350, or 525 mg eq.) on Week 17, 29, 41, and 53 as injection in deltoid muscle or gluteal muscle.
- Double Blind: Paliperidone Palmitate 1 Month Formulation: Participants received Paliperidone Palmitate 1-month formulation (PP1M) in a fixed dose that was administered at Week 9 at every month for 48 weeks, that is, participants received fixed dose injections of PP1M (50, 75, 100, or 150 mg eq.) as injection on deltoid muscle or gluteal muscle.
Arm/Group | Double Blind: Paliperidone Palmitate 3 Month Formulation | Double Blind: Paliperidone Palmitate 1 Month Formulation
Number analyzed (Participants) | 458 | 490
Percentage of Participants | 91.5 | 90.0

2. Secondary Outcome: Change From Double-Blind (DB) Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 48
Description: The neuropsychiatric symptoms of schizophrenia were assessed by means of the 30-item Positive and Negative Syndrome Scale (PANSS). The PANSS provides a total score (sum of the scores of all 30 items) ranging from 30 to 210, higher scores indicate more severe neuropsychiatric symptoms of schizophrenia. Scores for 3 subscales, that is, for positive subscale (sum of the scores of all 7 items) and negative subscale (sum of the scores of all 7 items) ranges from 7 (absent) to 49 (extreme psychopathology), and for the general psychopathology subscale (sum of the scores of all 16 items) score ranges from 16 (absent) to 112 (extreme psychopathology).
Time Frame: DB Baseline (Week 17) and 48 week or DB Endpoint
Population: mITT analysis set included all participants who were randomly assigned to treatment during Double-blind Phase, received at least 1 dose of study drug and did not have any errors in the delivery of active treatment. Here,N=number of participants analysed is the total participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind: Paliperidone Palmitate 3 Month Formulation | Double Blind: Paliperidone Palmitate 1 Month Formulation
Number analyzed (Participants) | 481 | 503
Units on a scale
  Baseline | 57.4 (8.56) | 58.1 (8.88)
  Change from Baseline at DB End point | -3.5 (12.50) | -4.3 (11.78)

3. Secondary Outcome: Change From DB Baseline in Clinical Global Impression Severity (CGI-S) Scale Score at Week 48
Description: The Clinical Global Impression Severity (CGI-S) rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: DB Baseline (Week 17) and 48 week or DB Endpoint
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind: Paliperidone Palmitate 3 Month Formulation | Double Blind: Paliperidone Palmitate 1 Month Formulation
Number analyzed (Participants) | 481 | 504
Units on a scale
  Baseline | 2.9 (0.57) | 2.9 (0.66)
  Change from Baseline at DB End point | -0.1 (0.84) | -0.1 (0.75)

4. Secondary Outcome: Change From DB Baseline in Personal and Social Performance (PSP) Total Score at Week 48
Description: The Personal and Social Performance (PSP) scale assesses degree of a participant's dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. Score ranges from 1 to 100. Participants with a score of 71 to 100 have mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision.
Time Frame: DB Baseline (Week 17) and 48 week or DB Endpoint
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind: Paliperidone Palmitate 3 Month Formulation | Double Blind: Paliperidone Palmitate 1 Month Formulation
Number analyzed (Participants) | 474 | 495
Units on a scale
  Baseline | 65.5 (10.40) | 65.0 (11.06)
  Change from Baseline at DB End point | 1.3 (10.22) | 1.9 (9.21)

5. Secondary Outcome: Percentage of Participants Who Met the Criteria for Symptomatic Remission Based on Andreasen Criteria
Description: Symptomatic remission criterion was defined as having a simultaneous score of mild or less on all selected PANSS items (P1, P2, P3, N1, N4, N6, G5, and G9). Symptomatic remission was defined for the last 6 months of the Double-blind Phase as meeting the remission criterion during the 6 months prior to the End of study visit during the Double-blind Phase, with one excursion allowed.
Time Frame: Weeks 41 to 65
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Double Blind: Paliperidone Palmitate 3 Month Formulation | Double Blind: Paliperidone Palmitate 1 Month Formulation
Number analyzed (Participants) | 483 | 512
Percentage of Participants | 58.4 [0.89 to 1.08] | 59.2 [0.89 to 1.08]

6. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Subscales Score at Week 48
Description: as for outcome 2
Time Frame: DB Baseline (Week 17) and 48 week or DB Endpoint
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind: Paliperidone Palmitate 3 Month Formulation | Double Blind: Paliperidone Palmitate 1 Month Formulation
Number analyzed (Participants) | 483 | 512
Units on a scale
  Positive subscale: Baseline | 11.9 (3.12) | 12.0 (3.19)
  Positive subscale:Change at Endpoint | -0.6 (4.31) | -0.9 (3.70)
  Negative subscale: Baseline | 17.3 (4.27) | 17.3 (4.11)
  Negative subscale:Change at Endpoint | -1.4 (3.63) | -1.4 (3.67)
  General psychopathology : Baseline | 28.2 (4.55) | 28.8 (4.79)
  General psychopathology : Change at Endpoint | -1.4 (6.77) | -2.0 (6.57)

7. Secondary Outcome: Change From Baseline in Marder Factor Subscale Score at Week 48
Description: 5 PANSS Marder factor scores (positive symptoms [range:8 to 56], negative symptoms [range: 7 to 49], disorganized thoughts [range: 7 to 49], uncontrolled hostility/excitement [range: 4 to 28], and anxiety/depression [range: 4 to 28]) were examined to gain insight into the symptoms affected by treatment with the study drug. Negative change from baseline in subscales score for positive symptoms, negative symptoms, disorganized thoughts, uncontrolled hostility/excitement, and anxiety/depression indicates improvement in various symptoms of schizophrenia.
Time Frame: DB Baseline (Week 17) and 48 week or DB Endpoint
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind: Paliperidone Palmitate 3 Month Formulation | Double Blind: Paliperidone Palmitate 1 Month Formulation
Number analyzed (Participants) | 483 | 512
Units on a scale
  Positive symptoms factor: Baseline | 15.7 (3.66) | 15.8 (3.88)
  Positive symptoms factor:Change at Endpoint | -1.1 (4.61) | -1.4 (4.16)
  Negative symptoms factor: Baseline | 16.2 (4.03) | 16.3 (3.90)
  Negative symptoms factor : Change at Endpoint | -1.4 (3.57) | -1.3 (3.80)
  Disorganized thoughts factor :Baseline | 14.2 (3.20) | 14.3 (3.17)
  Disorganized thoughts factor:Change at Endpoint | -1.2 (3.36) | -1.2 (3.24)
  Uncontrolled hostility Factor:Baseline | 5.2 (1.64) | 5.4 (1.77)
  Uncontrolled hostility Factor:Change at Endpoint | 0.2 (2.31) | -0.2 (2.21)
  Anxiety/depression factor:Baseline | 6.1 (2.02) | 6.3 (2.12)
  Anxiety/depression factor:Change at Endpoint | -0.0 (2.69) | -0.2 (2.43)

ADVERSE EVENTS:
Time Frame: From signing of informed consent form up to Follow-Up Visit (4 or 12 Weeks after study drug administration)
Description: For Double-blind (DB) phase, safety analysis set included all participants who were randomly assigned to treatment during DB Phase and received at least 1 dose of DB study drug. For Open-label Phase, all participants who received at least 1 dose of open-label study drug and were included in summary of safety assessments for that phase.
Arm/Group | Open-Label: Paliperidone Palmitate (PP1M) 1-month Formulation | Double-Blind: Paliperidone Palmitate(PP3M) 3-month Formulation | Double-Blind: Paliperidone Palmitate(PP1M) 1-month Formulation
Serious Adverse Events (participants affected / at risk) | 101/1429 | 26/504 | 37/512
Other Adverse Events (participants affected / at risk) | 457/1429 | 212/504 | 208/512
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label: Paliperidone Palmitate (PP1M) 1-month Formulation (N=1429) | Double-Blind: Paliperidone Palmitate(PP3M) 3-month Formulation (N=504) | Double-Blind: Paliperidone Palmitate(PP1M) 1-month Formulation (N=512)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 1
Drug Ineffective (General disorders) | 2 | 0 | 0
Drug Withdrawal Syndrome (General disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Meningitis Bacterial (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 0 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Akathisia (Nervous system disorders) | 4 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Stupor (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Acute Psychosis (Psychiatric disorders) | 2 | 0 | 0
Adjustment Disorder (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1
Alcohol Abuse (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 0 | 2
Anxiety Disorder (Psychiatric disorders) | 2 | 1 | 0
Delusion (Psychiatric disorders) | 4 | 1 | 2
Depressed Mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1
Hallucination, Auditory (Psychiatric disorders) | 6 | 1 | 0
Hostility (Psychiatric disorders) | 1 | 0 | 0
Hypomania (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Irritability (Psychiatric disorders) | 3 | 0 | 0
Neurosis (Psychiatric disorders) | 1 | 0 | 0
Persecutory Delusion (Psychiatric disorders) | 1 | 0 | 1
Psychiatric Symptom (Psychiatric disorders) | 4 | 2 | 2
Psychotic Disorder (Psychiatric disorders) | 14 | 1 | 2
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 31 | 12 | 11
Schizophrenia, Paranoid Type (Psychiatric disorders) | 0 | 0 | 2
Self Injurious Behaviour (Psychiatric disorders) | 1 | 0 | 0
Substance-Induced Psychotic Disorder (Psychiatric disorders) | 2 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 6 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 3 | 0 | 4
Tension (Psychiatric disorders) | 1 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 1
Menstrual Disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label: Paliperidone Palmitate (PP1M) 1-month Formulation (N=1429) | Double-Blind: Paliperidone Palmitate(PP3M) 3-month Formulation (N=504) | Double-Blind: Paliperidone Palmitate(PP1M) 1-month Formulation (N=512)
Injection Site Induration (General disorders) | 40 | 14 | 6
Injection Site Pain (General disorders) | 127 | 12 | 14
Nasopharyngitis (Infections and infestations) | 66 | 36 | 33
Weight Decreased (Investigations) | 10 | 14 | 14
Weight Increased (Investigations) | 64 | 105 | 109
Akathisia (Nervous system disorders) | 78 | 20 | 14
Headache (Nervous system disorders) | 46 | 18 | 26
Anxiety (Psychiatric disorders) | 79 | 27 | 22
Insomnia (Psychiatric disorders) | 94 | 16 | 24
Hypertension (Vascular disorders) | 11 | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.